CLINICAL TRIAL: NCT01923805
Title: A Prospective Randomized Evaluation of a Collagen/Thrombin Autologous Platelet Hemostatic Agent During Revision Knee Arthroplasty
Brief Title: Vitagel Revision Total Knee Arthroplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty enrolling patients
Sponsor: The Cleveland Clinic (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-1128
Record Dates: First submitted 2013-07-26; First posted 2013-08-16 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: Failed Total Knee Arthroplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Experimental): Vitagel
  Interventions: Device: Vitagel
- Control (No Intervention): Standard of care for surgical hemostasis.

INTERVENTIONS:
Device: Vitagel — Vitagel
  Arms: Treatment Group

SUMMARY:
This prospective study will evaluate the effectiveness of Vitagel (VG) in reducing blood loss associated with Revision Total Knee Arthroplasty (RTKA) procedures by assessing the patient's change in hemoglobin/hematocrit. Transfusion rates with the use of VG compared to the current standard of care will also be evaluated. The effectiveness of VG to potentially reduce pain, and increase return to function and quality of life will be assessed through the modified Knee Injury and Osteoarthritis Outcome Score (Modified KOOS), the Numerical Assessment Pain Scale (NAPS), and the SF-12 health survey. Analgesic use will be recorded post-operatively.

DETAILED DESCRIPTION:
This is a prospective, randomized, blinded clinical trial involving 4 orthopedic surgeons who perform Revision Total Knee Arthroplasty (RTKA), including Trevor Murray (PI), Viktor Krebs, Robert Molloy, and Carlos Higuera. A total of eighty subjects scheduled for RTKA, who meet all inclusion criteria and exhibit none of the exclusion criteria will be invited to participate in the study. Only subjects who sign the Institutional Review Board-approved Informed Consent Form will be entered into the Study.

In the forty treatment Subjects, VG will be applied to each surgical site. The forty control subjects will receive the surgeon's standard of care, without the use of any other hemostatic agents. The subjects will not be informed of their assignment, and the research investigator making the determination on blood transfusion requirements for all study subjects will also be blinded to the subject assigned arm of the study. The research investigator performing RTKA will remain blinded to the study arm until the randomization envelope is opened, which will take place during surgery, after hemostasis is achieved using bovie electrocautery, and prior to closure of the knee capsule.

Assessments will be made per the Time and Events Schedule.

Subjects will be evaluated for intra- and post-operative complications, and all such events, should they occur, will be recorded during the course of the study. Details describing the event, cause of event, its treatment and resolution will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria in order to be considered appropriate candidates for participation in the study:

  1. Is scheduled for RTKA (may be the second stage/reimplantation of a two-stage revision for infection);
  2. Is able and willing to provide voluntary written informed consent for participation in the study and able to comply with protocol requirements;
  3. Is between the ages of 18 and 85 at the time of surgery. Both male and female will be included;
  4. Is physically and mentally willing and able to comply with the clinical and evaluation follow-up schedule;

Exclusion Criteria:

* The following exclusion criteria address safety and follow-up concerns or contraindications that could confound the study. If a patient exhibits any one of the following criteria, the patient is not eligible to participate in this study:

  1. Is known to be sensitive to any materials of bovine origin;
  2. Is undergoing a bilateral RTKA;
  3. Is undergoing a single component revision (i.e. tibial or femoral component only)
  4. Is undergoing a polyethylene revision only
  5. Is predonating autologous blood;
  6. Have a preoperative platelet count of less than 100,000
  7. Have a previous history of venous thromboembolism or deep vein thrombosis;
  8. Have a medical condition requiring anticoagulation
  9. Currently using Coumadin;
  10. Have a history of Heparin induced thrombocytopenia or Lovenox induced thrombocytopenia;
  11. Have a history of rheumatoid arthritis or inflammatory arthritis;
  12. Have peripheral vascular disease;
  13. Have evidence of bleeding or metabolic-based hemolytic disorder (hemophilia or anticoagulation use), or hypercoaguable disorder;
  14. Have a history of liver disease. Patients with liver dysfunction from cirrhosis or hepatitis may have impaired production of factors in the clotting cascade which may make these individuals more prone to bleed, especially with the use of anticoagulants. For this reason, these patients will also be excluded from the study if a baseline INR is greater than 1.3 or APTT greater than 32.4;
  15. Have a history of failed treatment for abuse of, or are actively abusing, illegal drugs, solvents, or alcohol;
  16. Have a systemic infection or infection at site of surgery;
  17. Is a prisoner;
  18. Is pregnant or nursing and;
  19. Have a condition deemed by physician or medical staff to be non-conducive to patient's ability to complete the study, or a potential risk to the patient's health and well-being.

Exclusion Criteria (Intra-operative)

1. Clinical evidence of cancer and/or infection at surgical site
2. Use during the procedure of any other approved or unapproved product for the purpose of hemostasis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trevor Murray, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Study terminated early

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group | Control
Started (early termination) | 3 (early termination) | 5 (early termination)
Completed | 0 | 0
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Continuous [Mean (Full Range); unit: years] | 64 [59 to 69] | 57.8 [48 to 66] | 60.1 [48 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Transfusion Requirements
Description: The primary objective of this study is to test for significant differences in transfusion requirements in patients managed with RTKA.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 12 weeks.
Population: Data were not collected from participants enrolled in the study
Arm/Group | Treatment Group | Control
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

ADVERSE EVENTS:
Arm/Group | Treatment Group | Control
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/5
Other Adverse Events (participants affected / at risk) | 0/3 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=3) | Control (N=5)
Pulmonary Embolism, bilateral lower extremity deep vein thrombosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No